CLINICAL TRIAL: NCT05571722
Title: Linezolid or Vancomycin Surgical Site Infection Prophylaxis
Acronym: LOVip
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCAPHM22_0233
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Antibiotic Prophylaxis; General Surgery
MeSH Terms: interventions — Vancomycin; Linezolid

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The treatment scheme of the study does not allow for double-blinded manipulations. Postoperative evaluations and measurements will be performed in a blinded fashion by an investigator different from the physician who managed the patient in the operating room: SSI rates, adverse events, and length of stay. Statistical analyses will be performed in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Vancomycin (Active Comparator): Patients receive a dose of 30 mg/kg of vancomycin (2 hours infusion) starting 2.5 hours before the scheduled time of surgical incision as defined in the French guidelines.
  Interventions: Drug: Vancomycin Injection
- Experimental group: linezolid (Experimental): Patients receive a dose of 1200 mg of linezolid (30 minutes infusion) 30 minutes before the scheduled time of surgical incision.
  Interventions: Drug: Linezolid Injection

INTERVENTIONS:
Drug: Vancomycin Injection — Patients receive a dose of 30 mg/kg of vancomycin (2 hours infusion) starting 2.5 hours before the scheduled time of surgical incision as defined in the French guidelines.
  Arms: Control group: Vancomycin
Drug: Linezolid Injection — Patients receive a dose of 1200 mg of linezolid (30 minutes infusion) 30 minutes before the scheduled time of surgical incision.
  Arms: Experimental group: linezolid

SUMMARY:
Anesthesia and surgical guidelines recommend the administration of a surgical antibiotic prophylaxis for patients undergoing "clean" surgery. The prescribed antibiotic should target the bacteria most commonly found in surgical site infections (SSIs) and the duration of administration should not exceed 24 hours to minimize the ecological risk of bacterial resistance emergence. Guidelines provide a framework for the administration of surgical antibiotic prophylaxis but their effectiveness is regularly re-evaluated by measuring the rates of SSIs and the microorganisms responsible for infectious complications after surgery.

The majority of interventions required the use of first or second generation cephalosporins as surgical antibiotic prophylaxis. For patients with allergy to beta-lactams, clindamycin and vancomycin are proposed as alternatives. In the patients with methicillin-resistant S. aureus (MRSA) colonization or if those at risk of developing MRSA-associated SSI (hospital ecology, previous antibiotic treatment), only vancomycin is recommended. Vancomycin pharmacokinetics and pharmacodynamics is complex and its tissue absorption varies according to the level of tissue inflammation. This is a difficult molecule to handle, exclusively administered via intravenous route.

Linezolid is a synthetic antibiotic from the oxazolidinone class. By binding to the rRNA on the 30S and 50S ribosomal subunits, it inhibits the bacterial synthesis. It is therefore a bacteriostatic antibiotic approved for the treatment of both methicillin susceptible S. aureus (MSSA) and MRSA infections. It also covers a broad spectrum of Gram positive bacteria. Its pharmacokinetics allows rapid intravenous infusion, with rapid penetration into bone and soft tissue of the surgical site during hip surgery. A large Cochrane meta-analysis reported that linezolid was superior to vancomycin in skin infections, including MRSA infections, albeit with low quality evidence.

We therefore hypothesized that linezolid can be used instead of vancomycin for beta-lactam allergic patients and patients at risk of MRSA-associated SSI in general surgery.

DETAILED DESCRIPTION:
Anesthesia and surgical guidelines recommend the administration of a surgical antibiotic prophylaxis for patients undergoing "clean" surgery. The prescribed antibiotic should target the bacteria most commonly found in surgical site infections (SSIs) and the duration of administration should not exceed 24 hours to minimize the ecological risk of bacterial resistance emergence.

Surgical site infections are devastating complications occurring after surgery. They can lead to prolonged and burdensome duration of hospitalization, resulting in impaired outcomes and additional costs.

Many infections are associated with Gram positive bacteria, mainly Staphylococcus aureus and Staphylococcus spp with negative coagulase. Large European cohorts reported that less than 10% of SSIs were associated with Gram negative bacteria, justifying the use of 1st and 2nd generation cephalosporin, clindamycin and vancomycin as surgical antibiotic prophylaxis.

Guidelines provide a framework for the administration of surgical antibiotic prophylaxis but protocols are discussed at the local level with an agreement between surgeons, anesthesiologists, infectious diseases specialists, microbiologists and pharmacists. They are subject to economic analyses, including head-to-head comparisons of different options. Their effectiveness is regularly re-evaluated by measuring the rates of SSIs and the microorganisms responsible for infectious complications after surgery.

The majority of interventions required the use of first or second generation cephalosporins as surgical antibiotic prophylaxis. For patients with allergy to beta-lactams, clindamycin and vancomycin are proposed as alternatives. In the patients with methicillin-resistant S. aureus (MRSA) colonization or if those at risk of developing MRSA-associated SSI (hospital ecology, previous antibiotic treatment), only vancomycin is recommended. Actually, clindamycin was found to be less effective than beta-lactams or vancomycin in reducing the risk of SSI; the reported odds ratios (OR) for SSIs as compared to cefazolin range from an OR of 1.38 (95%CI 1.11 to 1.71) to OR 3.45 (95% CI 1.84 to 6.47).

Vancomycin is a large glycopeptide molecule, effective against a wide variety of Gram positive bacteria. The pharmacokinetics and pharmacodynamics (PK/PD) of vancomycin is complex, involving multicompartmental models. Its tissue absorption varies according to the level of tissue inflammation. It is exclusively administered via intravenous route. This is a difficult molecule to handle: specific international guidelines for its management have been published. In surgical antibiotic prophylaxis, French guidelines recommend a single loading dose infusion of vancomycin. It is recommended that loading doses of vancomycin should be administered as a low-rate infusion to mitigate infusion-related adverse events such as red-man syndrome (rate of 10-15 mg/min representing ≥1 hour for 1000 mg). Despite decades of use, vancomycin dosing regimens are still debated. Vancomycin dosing is commonly based on the actual patient body weight, although the volume of distribution of vancomycin is not proportional to weight. Therefore, as loading dose should lead to a rapid attainment of therapeutic concentrations, high doses (30 mg/kg) have been proposed for surgical antibiotic prophylaxis with a capping threshold of 2000 mg to avoid overdosing and risk of acute renal failure. These doses rapidly achieve the area under the curve (AUC) over the minimal inhibitory concentration (MIC) (AUC/MIC) targets, assuming a MIC ≤1mg/L for MRSA. Such high doses require prolonged infused time (at least two hours) and the administration should be terminated 30 minutes prior to surgery. This recommendation can lead to suboptimal administration times, delays in surgery and may also preclude the use of vancomycin in outpatient surgery. A U.S cohort reported that vancomycin was administered in 64% of cases outside national and institutional standards and incomplete administration of vancomycin has been associated with higher rates of SSI. Furthermore, in a nationwide US sample published, half of the patients receiving vancomycin were underdosed, which was associated with an increased risk of SSI.

Linezolid is a synthetic antibiotic from the oxazolidinone class. By binding to the rRNA on the 30S and 50S ribosomal subunits, it inhibits the bacterial synthesis. It is therefore a bacteriostatic antibiotic approved for the treatment of both methicillin susceptible S. aureus (MSSA) and MRSA infections. It also covers a broad spectrum of Gram positive bacteria. Its pharmacokinetics allows rapid intravenous infusion, with achievement of peak plasma concentrations within 30 minutes. Linezolid has also been shown to penetrate rapidly into bone and soft tissue of the surgical site during hip surgery. A large Cochrane meta-analysis reported that linezolid was superior to vancomycin in skin infections, including MRSA infections, albeit with low quality evidence.

We therefore hypothesized that linezolid can be used instead of vancomycin for beta-lactam allergic patients and patients at risk of MRSA-associated SSI in general surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing any elective surgery for which vancomycin is recommended in the guidelines as an alternative to beta-lactams including: neurosurgery, cardiac surgery, orthopedic surgery, vascular surgery, penile and testicular surgery, gastric banding procedure in digestive surgery.

This inclusion criteria can lead to the inclusion of patients who undergo a re-intervention provided that the re-intervention is not due to a suspected or proven infection and that the patient was not included in LOVip at the time of his/her first intervention;

* Age ≥ 18 years-old;
* Known allergy to beta-lactams AND/OR suspected or proven MRSA colonization. Proven MRSA colonization is defined as a positive patient sample (any type of swab or biological fluid) for MRSA within 3 months prior to surgery. MRSA colonization is suspected when the patient undergoing surgery has received antibiotic treatment within 3 months prior to surgery or is undergoing re-intervention more than 5 days after the first surgery. MRSA is defined as a strain of Staphylococcus aureus resistant to oxacillin or cefoxitin, predicting non-susceptibility to all classes of beta-lactam antimicrobials (except anti-MRSA cephalosporins) (6). In contrast, MSSA is defined as an oxacillin sensitive strain of Staphylococcus aureus;
* Informed consent of the patient;
* Affiliated to a social security system or equivalent.

Exclusion Criteria:

* Surgery for suspected or proven SSI (definition of SSI provided on chapter 3.6.1 Primary endpoint as defined by (5, 7)) according to international definitions;
* Obesity defined by a body mass index (BMI) > 35 kg/m2 or a body weight > 100 kg;
* Chronic kidney disease defined as glomerular filtration rate (GFR) < 60 ml/min per 1.73m2;
* Known allergy to linezolid or vancomycin;
* Hematologic malignancy;
* Declared pregnancy or breastfeeding;
* Patient under legal protection regime for adults;
* Patient denying consent;
* Patient already included in LOVip for a previous surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1160 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2028-12-03 (Estimated); Study Completion 2029-12-03 (Estimated)

PRIMARY OUTCOMES:
Comparaison of the rates of SSIs in patients receiving vancomycin 30 mg/kg versus patients receiving linezolid 1200 mg as surgical antibiotic prophylaxis for all types of surgery | Day 30 after surgery
  The SSIs are defined according to the standardized and validated Centers for Disease Control (CDC) criteria, including three levels of infection (superficial, deep, organ or space) (10). These definitions were endorsed by Santé Publique France and are used by the ISO-Raisin Network for the surveillance of nosocomial infections.

SECONDARY OUTCOMES:
Assessment of SSIs rates in all patients after 365 days | 365 after surgery
  SSI rate following the same definitions as detailed in the primary endpoint
Comparaison of treatment compliance | Day-365
  Occurrence of one of the following items indicates 'non-compliance' with treatment (the other cases will be defined as 'compliance'):
  * Need for antibiotic treatment interruption
  * Dose of antibiotic effectively delivered to the patient prior to surgical incision <30 mg/kg for the vancomycin group or <1200 mg for the linezolid group
  * Time between antibiotic administration completion and surgical incision <30 minutes
  * Scheduled time of surgery postponed due to antibiotic administration
  * Rates of vancomycin infusion duration <2 hour
  * Rates of linezolid infusion duration <30 minutes
Number of days from hospital admission to surgery, from surgery to discharge, from inclusion to discharge | Day-365
Mortality rates In-hospital, at day-30, at day-90 and at day-365; | day-30, at day-90 and at day-365
Antibiotic-free days during the 30-days following surgery | Day-30
Rates of Gram positive and Gram negative infections of any sites requiring antibiotic treatments | Day-365
Rates of MSSA and MRSA infections | Day-365
Preference-based utility score | Day-365
  EuroQol five-level (EQ5D-5L) questionnaire and scale (assessed through a phone call at day-30), it is a score with 5 items rated from 0 to 100) measured in all patients (EQ5D-5L questionnaire, EQ5D-5L scale)
Total costs of care during the 30-day study period and associated costs over the 365-day study period in all patients; | 30-Day and 365-day

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Anesthésie Réanimation - Hôpital Nord (AP-HM), Marseille, France

IPD SHARING:
Plan to Share IPD: No